CLINICAL TRIAL: NCT00177034
Title: Characterization of Keratinocyte Populations From Normal, Perilesional and Lesional Skin in Vitiligo Patients by Laser Capture Microdissection and Gene Array Analysis Before and After Narrow Band UVB Treatment
Brief Title: Examination Of Vitiligo Skin Samples Before and After UVB Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Mimi Cho, MD (Individual)
Collaborators: American Skin Association (Other)
Responsible Party: Sponsor
Organization: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0310M52823
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Vitiligo
Keywords: Keratinocyte
MeSH Terms: conditions — Vitiligo

INTERVENTIONS:
Drug: Narrow Band UVB Treatment

SUMMARY:
The keratinocytes of lesional skin of vitiligo compared to normal and perilesional skin will differentially express genes correlating with melanocyte death. Narrow Band UVB should then hopefully reverse the pattern of gene expression back toward normal.

DETAILED DESCRIPTION:
Vitiligo is a disease caused by the disappearance of melanocytes in the epidermis. The pathogenesis of vitiligo is multifactorial. Theories include autoimmunity, neural, apoptosis and cytotoxicity. The medical treatments for vitiligo are marginal with a 40-60% response rate which does not guarantee full repigmentation. Understanding the pathogenesis of vitiligo will allow better targets for treatment.

Previous analysis of skin biopsies have found several of the changes in gene expression occurred in immune regulation, DNA replication and repair, oncogenes, signal transducers and transcription factors. These results give us insight as to what happens in lesional vs nonlesional skin which contains the epidermis, dermis, fat, blood vessels and immune cells.

We have the technology today to study specific cell populations from tissue by the use of laser capture microdissection. We propose to use this technique to study the keratinocyte population in vitiligo skin because past evidence suggests that they may play a role. In addition, the role keratinocytes in vitiligo may be important for treatment as this would be the ideal target for therapy. Keratinocytes have been studied in vitiligo.

The aim of the study is to isolate keratinocytes from normal skin, perilesional and lesional skin in vitiligo patients by laser capture microdissection and characterize their gene expression profile by gene microarray analysis and to compare keratinocyte gene expression in normal, perilesional and lesional vitiligo skin before and after narrow band UVB treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients should have non-treated symmetrically active vitiligo for 3 months.

Exclusion Criteria:

Less than 18 years old and older that 65, pregnant women, segmental or nonactive vitiligo, patients treated for vitiligo in past 3 month, patients on topical steroid medications, topical tacrolimus or elidel, patients receiving ultraviolet therapy including narrow band UVB, PUVA or tanning beds.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2004-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Once genes profiling in keratinocytes between lesional and nonlesional skin is accomplished, we would like to characterize these keratinocyte populations after therapy.

SECONDARY OUTCOMES:
Keratinocytes have not been studied by gene expression analysis in this setting. The results from microarray analysis will be useful to see if the difference between lesional and nonlesional gene expression is reversed by therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Cho, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States